CLINICAL TRIAL: NCT05180188
Title: A Clinical Trial, Investigating the Effect of a Home-based Moderate Intensity Training Program on Oxidative Capacity and Hemodynamics in Patients With Truncating Genetic Variants in TTN.
Brief Title: Moderate Intensity Training in Patients With Truncating Genetic Variants in TTN.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ida Finsen Flensted, Bach.med., Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 75682
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Cardiomyopathies; Truncation Mutation; TTN
Keywords: TTNtv mutation; Intensity training; Exercise; VO2 max; Cardiac output
MeSH Terms: conditions — Cardiomyopathies; Motor Activity

STUDY DESIGN:
Intervention Model Description: The crossover trial has a two-period design. In the first study period, participants will not be exposed to any intervention and will be advised to not start any new medications, diets or participate in any activities which could influence their health. In the second period, participants will perform regular moderate-intensity exercise 3 times/week. Both study periods will last 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo periode (No Intervention): In the first study period, participants will not be exposed to any intervention and will be advised to not start any new medications, diets or participate in any activities which could influence their health.
- Exercise periode (Experimental): In the second period, participants will perform regular moderate-intensity exercise 3 times/week.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training — In the 8-week training period, participants will have three training sessions with a duration of 30 minutes at 70% of VO2peak per week.
  Arms: Exercise periode

SUMMARY:
The aim is to investigate the effect of an 8-week moderate-intensity exercise program on aerobic fitness and cardiac contractility in patients with truncations of the sarcomeric protein titin.

DETAILED DESCRIPTION:
Mutations leading to truncations of the large sarcomeric protein titin was discovered in 2012 as the most prevalent genetic cause of familial dilated cardiomyopathy, affecting approximately 25% of all cases of familial dilated cardiomyopathy. The dilated cardiomyopathy phenotype associated with truncating titin variants (TTNtv) is associated with a high prevalence of arrhythmias but is generally thought to represent a relatively mild DCM phenotype, which often responds well to medical therapy.

In vitro experiments on human induced pluripotent stem cells show that TTNtv leads to sarcomere insufficiency, impaired responses to mechanical and β-adrenergic stress, and attenuated growth factor and cell signaling activation. Experiments in animal models suggest patients with TTNtv are intolerant to long-lasting hemodynamic stress. This finding is supported by clinical studies in which a significant proportion of patients with peripartum cardiomyopathy, alcoholic cardiomyopathy and chemotherapy-induced cardiomyopathy were found to carry TTNtv.

So far, no interventional studies have been carried out specifically in patients with TTNtv. In an older study putative variants in TTN have been suggested to be associated with cardiac adaptations to endurance training, namely the rate of change in stroke volume during submaximal exercise.

Previous interventional exercise-studies in patients with a range of mutations in genes encoding proteins of the cytoskeleton, sarcomere, ion-channels and enzymes of the mitochondrial respiratory chain, safely improves oxidative fitness. Studies carried out on patients with heart failure of mixed etiologies and in patients with hypertrophic cardiomyopathy reveals similar beneficial effects of exercise. These studies reject the idea that training "diseased" muscle tissue leads to further muscle damage or is ineffective.

Many patients with cardiomyopathy often lead a sedentary life but aspire to live a physically active lifestyle and take advantage of the many documented health benefits of exercise. However, recommendations for engaging in physical activity in patients with heart failure and cardiomyopathies are vague since proper evidence does not exist for each genetic disorder.

In large-scale, prospective studies, it has been shown that physical fitness level and all-cause mortality are inversely related, even when corrected for other known risk factors. VO2peak reflects the physiological correlate of oxidative capacity in the muscular and cardiovascular systems. Low VO2peak is linked with an increased risk of ischemic heart disease, cancer and metabolic syndrome.

As a result, increasing VO2peak in patients with cardiomyopathy, who often have low baseline values of VO2peak, could lead to substantial long-term health benefits.

The study is an open label, non-randomized clinical crossover trial, investigating the effect of an 8-week exercise program in patients with pathogenic TTN variants that dispose or has resulted in cardiomyopathy.

The crossover trial has a two-period design. In the first study period, participants will not be exposed to any intervention and will be advised to not start any new medications, diets or participate in any activities which could influence their health. In the second period, participants will perform regular moderate-intensity exercise 3 times/week. Both study periods will last 8 weeks.

Based on results from prior trials we estimated that training would improve VO2peak by 10% (an estimated absolute increase of 2.5 ml O2/kg/min) with a standard deviation of 8.5%. Accordingly, we estimated that inclusion of 10 subjects would provide a power of 91% to detect this difference at a significance level of 0.05, using a paired t-test. Assuming a drop-out-rate of 20% a total of 14 patients should as a minimum be enrolled in the study. As a result, we aimed for the inclusion of a minimum of 14 trial participants, but up to 27 (if practically feasible) to make the evaluation of underlying physiological mechanisms leading to improved fitness possible.

Our hypothesis is that moderate-intensity exercise training safely improves oxidative capacity and that beneficial effects are partly caused by improvements in cardiac contractility.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Mutations in the TTN gene leading to truncating variants in cardiac expressed exons of titin.
3. A clinical diagnosis of dilated cardiomyopathy or fulfulling criteria for the diagnosis of heart failure or hypokinetic non-dilated cardiomyopathy.

Exclusion Criteria:

1. New York Heart Association functional class IV.
2. Patients with a left ventricular assist device or who have had a heart transplant.
3. Change in heart failure medications within the last month.
4. CRT implantation within the last 6 months.
5. Inability to perform exercise due to orthopedic or other non-cardiovascular limitations.
6. Clinical history of exercise-induced syncope likely caused by ventricular tachyarrhythmias.
7. Current participation in moderate or high intensity exercise exceeding 2.5 hours/per week.
8. Inability to give informed consent.
9. Pregnant women.
10. Severe vascular disease (IE claudicatio intermittens).
11. Severe valvular disease (moderate aortic stenosis/regurgitation or severe mitral regurgitation/stenosis).
12. Life expectancy less than 12 months.
13. Expected reduced compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Difference in change in peak oxygen uptake (VO2peak) as measured in an incremental cycle-ergometer exercise test to exhaustion, in the placebo vs intervention period | 8 weeks
  The VO2peak will be defined as the 20 consecutive seconds with the highest average VO2 during the incremental cycle-ergometer exercise test to exhaustion.

SECONDARY OUTCOMES:
Difference in change in left ventricular stroke volume at approximately 50% of maximal exertion in the placebo vs intervention period. | 8 weeks
  Left ventricular stroke volume will be measured at the same load after the intervention periode and the placebo periode.
Change in blood volume with training. | 8 weeks
Change in hemoglobin mass with training. | 8 weeks
Difference in change in cardiac output at approximately 50% of maximal exertion in the placebo vs intervention period. | 8 weeks
  Cardiac output will be measured at the same load after the intervention periode and the placebo periode.
Difference in change in cardiac output at 100% of VO2peak, in the placebo vs intervention period. | 8 weeks
  The VO2peak will be defined as the 20 consecutive seconds with the highest average
Difference in change in left ventricular stroke volume at 100% of VO2peak, in the placebo vs intervention period. | 8 weeks
  The VO2peak will be defined as the 20 consecutive seconds with the highest average
Difference in change in cardiac index at rest and during exercise | 8 weeks
Global longitudinal strain as measured by echocardiography | 8 weeks
Left ventricular volumetric measures from 3D echocardiography | 8 weeks
Change in systemic blood pressure | 8 weeks
Maximal workload in the maximal exercise test | 8 weeks
Performance in a 6-minute walk test | 8 weeks
Quality of life indicators as measured in the Short Form Health Survey (SF-36) | 8 weeks
Changes in cardiac and skeletomuscular biomarkers (CKMB, CK, NT proBNP, myoglobin, TnT, TnI) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Vissing, MD PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen Neuromuscular Center, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herman DS, Lam L, Taylor MR, Wang L, Teekakirikul P, Christodoulou D, Conner L, DePalma SR, McDonough B, Sparks E, Teodorescu DL, Cirino AL, Banner NR, Pennell DJ, Graw S, Merlo M, Di Lenarda A, Sinagra G, Bos JM, Ackerman MJ, Mitchell RN, Murry CE, Lakdawala NK, Ho CY, Barton PJ, Cook SA, Mestroni L, Seidman JG, Seidman CE. Truncations of titin causing dilated cardiomyopathy. N Engl J Med. 2012 Feb 16;366(7):619-28. doi: 10.1056/NEJMoa1110186. PMID 22335739
- [Background] Tayal U, Prasad S, Cook SA. Genetics and genomics of dilated cardiomyopathy and systolic heart failure. Genome Med. 2017 Feb 22;9(1):20. doi: 10.1186/s13073-017-0410-8. PMID 28228157
- [Background] Ahlberg G, Refsgaard L, Lundegaard PR, Andreasen L, Ranthe MF, Linscheid N, Nielsen JB, Melbye M, Haunso S, Sajadieh A, Camp L, Olesen SP, Rasmussen S, Lundby A, Ellinor PT, Holst AG, Svendsen JH, Olesen MS. Rare truncating variants in the sarcomeric protein titin associate with familial and early-onset atrial fibrillation. Nat Commun. 2018 Oct 17;9(1):4316. doi: 10.1038/s41467-018-06618-y. PMID 30333491
- [Background] Corden B, Jarman J, Whiffin N, Tayal U, Buchan R, Sehmi J, Harper A, Midwinter W, Lascelles K, Markides V, Mason M, Baksi J, Pantazis A, Pennell DJ, Barton PJ, Prasad SK, Wong T, Cook SA, Ware JS. Association of Titin-Truncating Genetic Variants With Life-threatening Cardiac Arrhythmias in Patients With Dilated Cardiomyopathy and Implanted Defibrillators. JAMA Netw Open. 2019 Jun 5;2(6):e196520. doi: 10.1001/jamanetworkopen.2019.6520. PMID 31251381
- [Background] Tayal U, Newsome S, Buchan R, Whiffin N, Walsh R, Barton PJ, Ware JS, Cook SA, Prasad SK. Truncating Variants in Titin Independently Predict Early Arrhythmias in Patients With Dilated Cardiomyopathy. J Am Coll Cardiol. 2017 May 16;69(19):2466-2468. doi: 10.1016/j.jacc.2017.03.530. No abstract available. PMID 28494986
- [Background] Choi SH, Weng LC, Roselli C, Lin H, Haggerty CM, Shoemaker MB, Barnard J, Arking DE, Chasman DI, Albert CM, Chaffin M, Tucker NR, Smith JD, Gupta N, Gabriel S, Margolin L, Shea MA, Shaffer CM, Yoneda ZT, Boerwinkle E, Smith NL, Silverman EK, Redline S, Vasan RS, Burchard EG, Gogarten SM, Laurie C, Blackwell TW, Abecasis G, Carey DJ, Fornwalt BK, Smelser DT, Baras A, Dewey FE, Jaquish CE, Papanicolaou GJ, Sotoodehnia N, Van Wagoner DR, Psaty BM, Kathiresan S, Darbar D, Alonso A, Heckbert SR, Chung MK, Roden DM, Benjamin EJ, Murray MF, Lunetta KL, Lubitz SA, Ellinor PT; DiscovEHR study and the NHLBI Trans-Omics for Precision Medicine (TOPMed) Consortium. Association Between Titin Loss-of-Function Variants and Early-Onset Atrial Fibrillation. JAMA. 2018 Dec 11;320(22):2354-2364. doi: 10.1001/jama.2018.18179. PMID 30535219
- [Background] Verdonschot JAJ, Hazebroek MR, Derks KWJ, Barandiaran Aizpurua A, Merken JJ, Wang P, Bierau J, van den Wijngaard A, Schalla SM, Abdul Hamid MA, van Bilsen M, van Empel VPM, Knackstedt C, Brunner-La Rocca HP, Brunner HG, Krapels IPC, Heymans SRB. Titin cardiomyopathy leads to altered mitochondrial energetics, increased fibrosis and long-term life-threatening arrhythmias. Eur Heart J. 2018 Mar 7;39(10):864-873. doi: 10.1093/eurheartj/ehx808. PMID 29377983
- [Background] Roberts AM, Ware JS, Herman DS, Schafer S, Baksi J, Bick AG, Buchan RJ, Walsh R, John S, Wilkinson S, Mazzarotto F, Felkin LE, Gong S, MacArthur JA, Cunningham F, Flannick J, Gabriel SB, Altshuler DM, Macdonald PS, Heinig M, Keogh AM, Hayward CS, Banner NR, Pennell DJ, O'Regan DP, San TR, de Marvao A, Dawes TJ, Gulati A, Birks EJ, Yacoub MH, Radke M, Gotthardt M, Wilson JG, O'Donnell CJ, Prasad SK, Barton PJ, Fatkin D, Hubner N, Seidman JG, Seidman CE, Cook SA. Integrated allelic, transcriptional, and phenomic dissection of the cardiac effects of titin truncations in health and disease. Sci Transl Med. 2015 Jan 14;7(270):270ra6. doi: 10.1126/scitranslmed.3010134. PMID 25589632
- [Background] Jansweijer JA, Nieuwhof K, Russo F, Hoorntje ET, Jongbloed JD, Lekanne Deprez RH, Postma AV, Bronk M, van Rijsingen IA, de Haij S, Biagini E, van Haelst PL, van Wijngaarden J, van den Berg MP, Wilde AA, Mannens MM, de Boer RA, van Spaendonck-Zwarts KY, van Tintelen JP, Pinto YM. Truncating titin mutations are associated with a mild and treatable form of dilated cardiomyopathy. Eur J Heart Fail. 2017 Apr;19(4):512-521. doi: 10.1002/ejhf.673. Epub 2016 Nov 3. PMID 27813223
- [Background] Jansen M, Baas AF, van Spaendonck-Zwarts KY, Ummels AS, van den Wijngaard A, Jongbloed JDH, van Slegtenhorst MA, Lekanne Deprez RH, Wessels MW, Michels M, Houweling AC, Hoorntje ET, Helderman-van den Enden PJTM, Barge-Schaapveld DQCM, Peter van Tintelen J, van den Berg MP, Wilde AAM, Ploos van Amstel HK, Hennekam EAM, Asselbergs FW, Sijbrands EJG, Dooijes D. Mortality Risk Associated With Truncating Founder Mutations in Titin. Circ Genom Precis Med. 2019 May;12(5):e002436. doi: 10.1161/CIRCGEN.118.002436. PMID 31112426
- [Background] Verdonschot JAJ, Hazebroek MR, Wang P, Sanders-van Wijk S, Merken JJ, Adriaansen YA, van den Wijngaard A, Krapels IPC, Brunner-La Rocca HP, Brunner HG, Heymans SRB. Clinical Phenotype and Genotype Associations With Improvement in Left Ventricular Function in Dilated Cardiomyopathy. Circ Heart Fail. 2018 Nov;11(11):e005220. doi: 10.1161/CIRCHEARTFAILURE.118.005220. PMID 30571196
- [Background] Felkin LE, Walsh R, Ware JS, Yacoub MH, Birks EJ, Barton PJ, Cook SA. Recovery of Cardiac Function in Cardiomyopathy Caused by Titin Truncation. JAMA Cardiol. 2016 May 1;1(2):234-5. doi: 10.1001/jamacardio.2016.0208. No abstract available. PMID 27437901
- [Background] Hinson JT, Chopra A, Nafissi N, Polacheck WJ, Benson CC, Swist S, Gorham J, Yang L, Schafer S, Sheng CC, Haghighi A, Homsy J, Hubner N, Church G, Cook SA, Linke WA, Chen CS, Seidman JG, Seidman CE. HEART DISEASE. Titin mutations in iPS cells define sarcomere insufficiency as a cause of dilated cardiomyopathy. Science. 2015 Aug 28;349(6251):982-6. doi: 10.1126/science.aaa5458. PMID 26315439
- [Background] Huttner IG, Wang LW, Santiago CF, Horvat C, Johnson R, Cheng D, von Frieling-Salewsky M, Hillcoat K, Bemand TJ, Trivedi G, Braet F, Hesselson D, Alford K, Hayward CS, Seidman JG, Seidman CE, Feneley MP, Linke WA, Fatkin D. A-Band Titin Truncation in Zebrafish Causes Dilated Cardiomyopathy and Hemodynamic Stress Intolerance. Circ Genom Precis Med. 2018 Aug;11(8):e002135. doi: 10.1161/CIRCGEN.118.002135. PMID 30354343
- [Background] Gramlich M, Michely B, Krohne C, Heuser A, Erdmann B, Klaassen S, Hudson B, Magarin M, Kirchner F, Todiras M, Granzier H, Labeit S, Thierfelder L, Gerull B. Stress-induced dilated cardiomyopathy in a knock-in mouse model mimicking human titin-based disease. J Mol Cell Cardiol. 2009 Sep;47(3):352-8. doi: 10.1016/j.yjmcc.2009.04.014. Epub 2009 May 4. PMID 19406126
- [Background] Zhou Q, Kesteven S, Wu J, Aidery P, Gawaz M, Gramlich M, Feneley MP, Harvey RP. Pressure Overload by Transverse Aortic Constriction Induces Maladaptive Hypertrophy in a Titin-Truncated Mouse Model. Biomed Res Int. 2015;2015:163564. doi: 10.1155/2015/163564. Epub 2015 Oct 4. PMID 26504781
- [Background] Ware JS, Li J, Mazaika E, Yasso CM, DeSouza T, Cappola TP, Tsai EJ, Hilfiker-Kleiner D, Kamiya CA, Mazzarotto F, Cook SA, Halder I, Prasad SK, Pisarcik J, Hanley-Yanez K, Alharethi R, Damp J, Hsich E, Elkayam U, Sheppard R, Kealey A, Alexis J, Ramani G, Safirstein J, Boehmer J, Pauly DF, Wittstein IS, Thohan V, Zucker MJ, Liu P, Gorcsan J 3rd, McNamara DM, Seidman CE, Seidman JG, Arany Z; IMAC-2 and IPAC Investigators. Shared Genetic Predisposition in Peripartum and Dilated Cardiomyopathies. N Engl J Med. 2016 Jan 21;374(3):233-41. doi: 10.1056/NEJMoa1505517. Epub 2016 Jan 6. PMID 26735901
- [Background] Ware JS, Amor-Salamanca A, Tayal U, Govind R, Serrano I, Salazar-Mendiguchia J, Garcia-Pinilla JM, Pascual-Figal DA, Nunez J, Guzzo-Merello G, Gonzalez-Vioque E, Bardaji A, Manito N, Lopez-Garrido MA, Padron-Barthe L, Edwards E, Whiffin N, Walsh R, Buchan RJ, Midwinter W, Wilk A, Prasad S, Pantazis A, Baski J, O'Regan DP, Alonso-Pulpon L, Cook SA, Lara-Pezzi E, Barton PJ, Garcia-Pavia P. Genetic Etiology for Alcohol-Induced Cardiac Toxicity. J Am Coll Cardiol. 2018 May 22;71(20):2293-2302. doi: 10.1016/j.jacc.2018.03.462. PMID 29773157
- [Background] Linschoten M, Teske AJ, Baas AF, Vink A, Dooijes D, Baars HF, Asselbergs FW. Truncating Titin (TTN) Variants in Chemotherapy-Induced Cardiomyopathy. J Card Fail. 2017 Jun;23(6):476-479. doi: 10.1016/j.cardfail.2017.03.003. Epub 2017 Mar 14. PMID 28315399
- [Background] Rankinen T, Rice T, Boudreau A, Leon AS, Skinner JS, Wilmore JH, Rao DC, Bouchard C. Titin is a candidate gene for stroke volume response to endurance training: the HERITAGE Family Study. Physiol Genomics. 2003 Sep 29;15(1):27-33. doi: 10.1152/physiolgenomics.00147.2002. PMID 12865504
- [Background] Sveen ML, Jeppesen TD, Hauerslev S, Kober L, Krag TO, Vissing J. Endurance training improves fitness and strength in patients with Becker muscular dystrophy. Brain. 2008 Nov;131(Pt 11):2824-31. doi: 10.1093/brain/awn189. Epub 2008 Sep 6. PMID 18776212
- [Background] Jeppesen TD, Duno M, Schwartz M, Krag T, Rafiq J, Wibrand F, Vissing J. Short- and long-term effects of endurance training in patients with mitochondrial myopathy. Eur J Neurol. 2009 Dec;16(12):1336-9. doi: 10.1111/j.1468-1331.2009.02660.x. Epub 2009 May 27. PMID 19486129
- [Background] Sveen ML, Jeppesen TD, Hauerslev S, Krag TO, Vissing J. Endurance training: an effective and safe treatment for patients with LGMD2I. Neurology. 2007 Jan 2;68(1):59-61. doi: 10.1212/01.wnl.0000250358.32199.24. PMID 17200494
- [Background] Vissing CR, Preisler N, Husu E, Prahm KP, Vissing J. Aerobic training in patients with anoctamin 5 myopathy and hyperckemia. Muscle Nerve. 2014 Jul;50(1):119-23. doi: 10.1002/mus.24112. Epub 2014 May 5. PMID 24639367
- [Background] Andersen G, Heje K, Buch AE, Vissing J. High-intensity interval training in facioscapulohumeral muscular dystrophy type 1: a randomized clinical trial. J Neurol. 2017 Jun;264(6):1099-1106. doi: 10.1007/s00415-017-8497-9. Epub 2017 May 3. PMID 28470591
- [Background] Orngreen MC, Olsen DB, Vissing J. Aerobic training in patients with myotonic dystrophy type 1. Ann Neurol. 2005 May;57(5):754-7. doi: 10.1002/ana.20460. PMID 15852373
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Background] Saberi S, Wheeler M, Bragg-Gresham J, Hornsby W, Agarwal PP, Attili A, Concannon M, Dries AM, Shmargad Y, Salisbury H, Kumar S, Herrera JJ, Myers J, Helms AS, Ashley EA, Day SM. Effect of Moderate-Intensity Exercise Training on Peak Oxygen Consumption in Patients With Hypertrophic Cardiomyopathy: A Randomized Clinical Trial. JAMA. 2017 Apr 4;317(13):1349-1357. doi: 10.1001/jama.2017.2503. PMID 28306757
- [Background] Maron BJ, Chaitman BR, Ackerman MJ, Bayes de Luna A, Corrado D, Crosson JE, Deal BJ, Driscoll DJ, Estes NA 3rd, Araujo CG, Liang DH, Mitten MJ, Myerburg RJ, Pelliccia A, Thompson PD, Towbin JA, Van Camp SP; Working Groups of the American Heart Association Committee on Exercise, Cardiac Rehabilitation, and Prevention; Councils on Clinical Cardiology and Cardiovascular Disease in the Young. Recommendations for physical activity and recreational sports participation for young patients with genetic cardiovascular diseases. Circulation. 2004 Jun 8;109(22):2807-16. doi: 10.1161/01.CIR.0000128363.85581.E1. PMID 15184297
- [Background] Blair SN, Kohl HW 3rd, Paffenbarger RS Jr, Clark DG, Cooper KH, Gibbons LW. Physical fitness and all-cause mortality. A prospective study of healthy men and women. JAMA. 1989 Nov 3;262(17):2395-401. doi: 10.1001/jama.262.17.2395. PMID 2795824
- [Background] Sattelmair J, Pertman J, Ding EL, Kohl HW 3rd, Haskell W, Lee IM. Dose response between physical activity and risk of coronary heart disease: a meta-analysis. Circulation. 2011 Aug 16;124(7):789-95. doi: 10.1161/CIRCULATIONAHA.110.010710. Epub 2011 Aug 1. PMID 21810663
- [Background] Laukkanen JA, Zaccardi F, Khan H, Kurl S, Jae SY, Rauramaa R. Long-term Change in Cardiorespiratory Fitness and All-Cause Mortality: A Population-Based Follow-up Study. Mayo Clin Proc. 2016 Sep;91(9):1183-8. doi: 10.1016/j.mayocp.2016.05.014. Epub 2016 Jul 18. PMID 27444976
- [Background] Ekelund LG, Haskell WL, Johnson JL, Whaley FS, Criqui MH, Sheps DS. Physical fitness as a predictor of cardiovascular mortality in asymptomatic North American men. The Lipid Research Clinics Mortality Follow-up Study. N Engl J Med. 1988 Nov 24;319(21):1379-84. doi: 10.1056/NEJM198811243192104. PMID 3185648
- [Background] Paffenbarger RS Jr, Hyde RT, Wing AL, Lee IM, Jung DL, Kampert JB. The association of changes in physical-activity level and other lifestyle characteristics with mortality among men. N Engl J Med. 1993 Feb 25;328(8):538-45. doi: 10.1056/NEJM199302253280804. PMID 8426621
- [Derived] Flensted IF, Stemmerik MG, Skriver SV, Axelsen KH, Christensen AH, Lundby C, Bundgaard H, Vissing J, Vissing CR. Exercise training improves cardiovascular fitness in dilated cardiomyopathy caused by truncating titin variants. Heart. 2024 Nov 25;110(24):1416-1425. doi: 10.1136/heartjnl-2024-323995. PMID 39317439